CLINICAL TRIAL: NCT05469139
Title: Assessing Brain Injury Using Portable Magnetic Resonance Imaging in Patients With Extracorporeal Membrane Oxygenation
Brief Title: Assessing Brain Injury Using Portable Magnetic Resonance Imaging (MRI)
Acronym: SAFE MRI
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Hyperfine (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00285716
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Acute Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Portable MRI group: Patients on ECMO who undergo portable MRI to assess brain injury within 24-48 hours of ECMO initiation
  Interventions: Diagnostic Test: Portable MRI acquisition

INTERVENTIONS:
Diagnostic Test: Portable MRI acquisition — Patients on ECMO will undergo a portable MRI of the brain

SUMMARY:
This study aims to assess the feasibility of assessing acute brain injury using a portable low field MRI in patients on ECMO.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is a life-saving therapy increasingly used in patients with refractory cardiopulmonary failure. The Extracorporeal Life Support Organization (ELSO) registry recently reported a 58% survival rate among patients who receive ECMO support, showing a significant mortality benefit in patients who would have not survived without ECMO. However, acute brain injury (ABI) is common in patients with ECMO support and leads to devastating consequences with significant morbidity and mortality. The mortality increases more than two-fold when ABI is present for both venoarterial (VA) and venovenous (VV) ECMO patients. The poor prognosis of ABI and neurological complications would suggest potential benefit from stringent and possibly even protocolized neurological monitoring to prevent or minimize further harm. This is particularly important as recent evidence promotes extracorporeal cardiopulmonary resuscitation (ECPR) as a rescue therapy for patients suffering from cardiac arrest of potentially reversible etiology. As clinical experience accumulates and ECPR becomes more widely used, neurological monitoring for complications and prognostication will be imperative for optimizing patient outcomes.

Although standardized neurological monitoring improves the detection of ABI, timely diagnosis and management for ABI in patients with ECMO support is still challenging due to the difficulty, impracticality, and danger of transporting ECMO patients to a CT scanner. Often, ECMO patients are unable to be transported to radiology suites because of the patients' persistent cardiopulmonary instability with multiple vasopressor requirements. In addition, even if head CT is performed in these patients, it is limited by poor sensitivity for detecting acute ischemic brain injury. Early neuroimaging is a key neuromonitoring aspect in the clinical evaluation of ABI. However, conventional magnetic resonance imaging (MRI) systems operate at high magnetic field strengths (1.5-3T) that require strict, access-controlled environments. Thus, limited access to timely brain scan with images of sufficient quality remains a significant barrier to effectively monitoring the occurrence and progression of ABI in ECMO.

Recent advances in low-field and portable MRI technology have enabled the acquisition of clinically meaningful imaging in the presence of ferromagnetic materials. A very low magnetic field strength, 64 magnetization transfer (mT), approximately 1/23 the field strength of a conventional MRI) provides a 5 Gauss line (safety zone) that is only about 2.5 feet from the center of the scanner. In a previous report, researchers were able to demonstrate the feasibility of a low-field, portable MRI in complex clinical care settings, such as intensive care units, without any adverse events or complications. In addition to reduced projectile motion, the use of low-field MRI may mitigate other safety concerns associated with high-field MRI, such as peripheral nerve stimulation (from gradients), a radiofrequency absorption and heating and acoustic noise.

The objective of this study is to assess acute brain injury with low-field, portable MRI of brain in patients with ECMO support.

This study will use the Hyperfine portable MRI machine which has FDA 510(k) clearance and is intended for use in intensive care units. The investigators' hypothesis is that low-field, portable MRI can detect ABI in patients with ECMO support, which may decrease the morbidity of patients on ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and over
* Patient supported with extracorporeal membrane oxygenation support (ECMO)
* Legally authorized representative has provided written informed consent

Exclusion Criteria:

* Patient has a contraindication for MRI such as:
* Implants such as pacemaker, defibrillator, implanted insulin pump, deep brain stimulator, vagus nerve stimulator, cochlear implant, or programmable shunt
* MRI incompatible surgical hardware such as staples, screws. ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, cochlear implant
* artificial hearts or heart valves with steel parts
* metal fragments
* shrapnel
* tattoos near the eye
* permanent make-up
* steel implants
* or other irremovable ferromagnetic objects
* Patient weight is over 440 lbs (or 200kg)
* Patient has Intra Aortic Balloon Pump (IABP), Implanted Ventricular Assist Device (VAD), or Percutaneous Ventricular Assist Device
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients on extracorporeal membrane oxygenation support (ECMO)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Acute brain injury as assessed by head CT scan | 48 hours from ECMO initiation
  compare results of routinely performed head CT scans with results from a low field MRI to determine whether acute brain injury can be assessed using a low field MRI in patients with ECMO support.

SECONDARY OUTCOMES:
prevalence of early acute brain injury as assessed by MRI scan | 24 hours from ECMO initiation
  use interpretations of low field MRI scans to determine the prevalence of early acute brain injury of patients with ECMO support at 24 hours
Image Quality | 48 hours from ECMO initiation
  compare image quality of low field MRI scans with the image quality of routinely performed head CT scans to assess the image quality of MR images for infarcts and hemorrhages
Impact of early detection as assessed by MRI | 48 hours from ECMO initiation
  assess anticoagulation strategies following low field MRI to determine the impact of early detection of acute brain injury on anticoagulation strategy
Association of Transcranial doppler ultrasound with ischemic infarct | 48 hours from ECMO initiation
  measure transcranial doppler ultrasounds and correlate the findings with the results of low field MRI to assess for an association between Transcranial doppler ultrasound (TCD) microembolic signal (MES) and the presence of ischemic infarct on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Min Cho, DO, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Texas Health Science Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Clinical Study report will be available upon completion of the study analysis

REFERENCES:
- [Background] McCarthy FH, McDermott KM, Kini V, Gutsche JT, Wald JW, Xie D, Szeto WY, Bermudez CA, Atluri P, Acker MA, Desai ND. Trends in U.S. Extracorporeal Membrane Oxygenation Use and Outcomes: 2002-2012. Semin Thorac Cardiovasc Surg. 2015 Summer;27(2):81-8. doi: 10.1053/j.semtcvs.2015.07.005. Epub 2015 Jul 22. PMID 26686427
- [Background] Thiagarajan RR, Barbaro RP, Rycus PT, Mcmullan DM, Conrad SA, Fortenberry JD, Paden ML; ELSO member centers. Extracorporeal Life Support Organization Registry International Report 2016. ASAIO J. 2017 Jan/Feb;63(1):60-67. doi: 10.1097/MAT.0000000000000475. PMID 27984321
- [Background] Cho SM, Canner J, Caturegli G, Choi CW, Etchill E, Giuliano K, Chiarini G, Calligy K, Rycus P, Lorusso R, Kim BS, Sussman M, Suarez JI, Geocadin R, Bush EL, Ziai W, Whitman G. Risk Factors of Ischemic and Hemorrhagic Strokes During Venovenous Extracorporeal Membrane Oxygenation: Analysis of Data From the Extracorporeal Life Support Organization Registry. Crit Care Med. 2021 Jan 1;49(1):91-101. doi: 10.1097/CCM.0000000000004707. PMID 33148951
- [Background] Cho SM, Canner J, Chiarini G, Calligy K, Caturegli G, Rycus P, Barbaro RP, Tonna J, Lorusso R, Kilic A, Choi CW, Ziai W, Geocadin R, Whitman G. Modifiable Risk Factors and Mortality From Ischemic and Hemorrhagic Strokes in Patients Receiving Venoarterial Extracorporeal Membrane Oxygenation: Results From the Extracorporeal Life Support Organization Registry. Crit Care Med. 2020 Oct;48(10):e897-e905. doi: 10.1097/CCM.0000000000004498. PMID 32931195
- [Background] Brooks SC, Anderson ML, Bruder E, Daya MR, Gaffney A, Otto CW, Singer AJ, Thiagarajan RR, Travers AH. Part 6: Alternative Techniques and Ancillary Devices for Cardiopulmonary Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S436-43. doi: 10.1161/CIR.0000000000000260. No abstract available. PMID 26472994
- [Background] Cho SM, Ziai W, Mayasi Y, Gusdon AM, Creed J, Sharrock M, Stephens RS, Choi CW, Ritzl EK, Suarez J, Whitman G, Geocadin RG. Noninvasive Neurological Monitoring in Extracorporeal Membrane Oxygenation. ASAIO J. 2020 Apr;66(4):388-393. doi: 10.1097/MAT.0000000000001013. PMID 31045914
- [Background] Sheth KN, Mazurek MH, Yuen MM, Cahn BA, Shah JT, Ward A, Kim JA, Gilmore EJ, Falcone GJ, Petersen N, Gobeske KT, Kaddouh F, Hwang DY, Schindler J, Sansing L, Matouk C, Rothberg J, Sze G, Siner J, Rosen MS, Spudich S, Kimberly WT. Assessment of Brain Injury Using Portable, Low-Field Magnetic Resonance Imaging at the Bedside of Critically Ill Patients. JAMA Neurol. 2020 Sep 8;78(1):41-7. doi: 10.1001/jamaneurol.2020.3263. Online ahead of print. PMID 32897296
- [Background] Campbell-Washburn AE, Ramasawmy R, Restivo MC, Bhattacharya I, Basar B, Herzka DA, Hansen MS, Rogers T, Bandettini WP, McGuirt DR, Mancini C, Grodzki D, Schneider R, Majeed W, Bhat H, Xue H, Moss J, Malayeri AA, Jones EC, Koretsky AP, Kellman P, Chen MY, Lederman RJ, Balaban RS. Opportunities in Interventional and Diagnostic Imaging by Using High-Performance Low-Field-Strength MRI. Radiology. 2019 Nov;293(2):384-393. doi: 10.1148/radiol.2019190452. Epub 2019 Oct 1. PMID 31573398
- [Background] Formica D, Silvestri S. Biological effects of exposure to magnetic resonance imaging: an overview. Biomed Eng Online. 2004 Apr 22;3:11. doi: 10.1186/1475-925X-3-11. PMID 15104797
- [Background] Hartwig V, Giovannetti G, Vanello N, Lombardi M, Landini L, Simi S. Biological effects and safety in magnetic resonance imaging: a review. Int J Environ Res Public Health. 2009 Jun;6(6):1778-98. doi: 10.3390/ijerph6061778. Epub 2009 Jun 10. PMID 19578460
- [Background] Shellock FG, Crues JV. Aneurysm clips: assessment of magnetic field interaction associated with a 0.2-T extremity MR system. Radiology. 1998 Aug;208(2):407-9. doi: 10.1148/radiology.208.2.9680568.
- [Background] Alorainy IA, Albadr FB, Abujamea AH. Attitude towards MRI safety during pregnancy. Ann Saudi Med. 2006 Jul-Aug;26(4):306-9. doi: 10.5144/0256-4947.2006.306. No abstract available. PMID 16885635